CLINICAL TRIAL: NCT03126071
Title: A Phase II Study of Raltitrexed-based Chemotherapy Plus Bevacizumab in Retreated Patients With Advanced Colorectal Cancer
Brief Title: Raltitrexed-based Chemotherapy Plus Bevacizumab in Retreated Patients With Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Liangjun Zhu M.M., Ward Director of Internal Medicine, Jiangsu Cancer Institute & Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBACC
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Advanced Colorectal Cancer
MeSH Terms: interventions — raltitrexed; Irinotecan; Oxaliplatin; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Raltitrexed and Irinotecan（RALIRI） plus Bevacizumab(AVASTIN) (Experimental): Irinotecan:250mg/m2 iv,90min,d1, Raltitrexed:3.0mg/m2,iv,15min,d1, Bevacizumab:7.5mg/kg iv,30min,d1,q3w. Maintenance: Raltitrexed(3.0mg/m2,iv,15min,d1,q3w)+Bevacizumab(7.5 mg/kg q3w)
  Interventions: Drug: Raltitrexed; Drug: Irinotecan; Drug: Bevacizumab
- Raltitrexed and Oxaliplatin（RALOX） plus Bevacizumab(AVASTIN) (Experimental): Oxaliplatin:130mg/m2 iv,120min,d1, Raltitrexed:3.0mg/m2,iv,15min,d1, Bevacizumab:7.5mg/kg iv,30min,d1,q3w. Maintenance: Raltitrexed(3.0mg/m2,iv,15min,d1,q3w)+Bevacizumab(7.5 mg/kg q3w)
  Interventions: Drug: Raltitrexed; Drug: Oxaliplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Raltitrexed — Raltitrexed:3mg/m2,iv 15min,d1,q3w.
Drug: Irinotecan — Irinotecan:250mg/m2,iv 90min,d1,q3w.
  Arms: Raltitrexed and Irinotecan（RALIRI） plus Bevacizumab(AVASTIN)
Drug: Oxaliplatin — Oxaliplatin:130mg/m2,iv 120min,d1,q3w.
  Arms: Raltitrexed and Oxaliplatin（RALOX） plus Bevacizumab(AVASTIN)
Drug: Bevacizumab — Bevacizumab:75mg/kg,iv 30min,d1,q3w.
  Other Names: Avastin

SUMMARY:
The objective is to investigate the efficacy and safety of raltitrexed-based chemotherapy plus bevacizumab in the treatment of advanced colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years;
* histological and/or cytological confirmation of ACC;
* disease progression while on first-line palliative fluoropyrimidine-based chemotherapy or relapse within 6 months after adjuvant chemotherapy;
* at least one measurable objective tumor lesion by spiral CT examination, the maximum diameter ≥ 1cm（according to RECIST 1.1）
* ECOG performance status 0-1
* life expectancy of at least 3 months
* satisfactory main organ function，laboratory test must meet the following criteria: hemoglobin (HGB) ≥90g/L, neutrophil count（ANC） ≥1.5×109/L, platelet count（PLT） ≥80×109/L, Serum creatinine（CR）≤1.5 upper normal limitation (UNL)，total bilirubin (TBil) ≤1.5 upper normal limitation (UNL), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 UNL (For patients with liver metastasis, the AST/ALT must be ≤5.0 UNL), Alkaline phosphatase（ALP）≤3 UNL(For patients with liver metastasis, the ALP must be ≤5.0 UNL);
* written informed consent

Exclusion Criteria:

* prior exposure to raltitrexed;
* Clinically significant cardiovascular disease, for example symptomatic coronary artery disease, myocardial infarction (<=6 months before treatment start),congestive heart failure （New York Heart Association ，NYHA>= grade 3）,stroke or transient ischemic attack
* Accept kidney dialysis treatment now
* chronic enteropathy on unresolved bowel obstruction;
* previous malignant disease other than carcinoma in situ of the cervix or basal cell carcinoma of the skin;
* the UGT1A1 *28（7/7）*6（A/A） gene type;
* pregnant or lactated women;
* Unsuitable for the study or other chemotherapy determined by investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 months
  Progression Free Survival

SECONDARY OUTCOMES:
OS | 15 months
  Overall Survival
ORR | 36 months
  Objective Response Rate
DCR | 36 months
  Disease Control Rate
AEs | 36 months
  Percentage of participants experiencing grade 3-5 adverse events

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Jiangsu Cancer Institute & Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Li S, Li X, Zhu Q, Gao J, Zhu C, Zhu L. Raltitrexed Chemotherapy Regimen Plus Bevacizumab as Second-Line Treatment for Metastatic Colorectal Cancer: A Prospective Multicenter Phase II Trial. Cancer Control. 2024 Jan-Dec;31:10732748241275012. doi: 10.1177/10732748241275012. PMID 39286935